CLINICAL TRIAL: NCT01321060
Title: Management of Sterile Fluid Collections in Patients With Severe Acute Pancreatitis:a Randomized Controlled Trial
Brief Title: Fluid Collections Management in Severe Acute Pancreatitis
Acronym: FCMSAP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanjing University School of Medicine (Other)
Collaborators: Jinling Hospital, China (Other)
Responsible Party: Principal Investigator, Weiqin Li, Director of surgical ICU, Nanjing University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RIGS
Record Dates: First submitted 2011-03-22; First posted 2011-03-23 (Estimated); Last update posted 2012-06-19 (Estimated); Status verified 2011-01

CONDITIONS: Acute Pancreatitis; Acute Pancreatic Fluid Collection
Keywords: severe acute pancreatitis; acute fluid collection; catheter drainage; repeated aspiration
MeSH Terms: conditions — Pancreatitis | interventions — Conservative Treatment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Conservative treatment (Active Comparator): Conservative treatment group with only drugs.
  Interventions: Drug: Conservative treatment
- Continuous catheter drainage (Experimental): Once the diameter of the fluid collection is more than 6cm, continuous catheter drainage will be applied.
  Interventions: Procedure: Catheter drainage
- Repeated aspiration (Experimental): Once the diameter of the fluid collection is more than 6cm, aspiration is applied and draw the tube out immediately after aspiration.
  Interventions: Procedure: Aspiration

INTERVENTIONS:
Procedure: Aspiration
  Arms: Repeated aspiration
Procedure: Catheter drainage
  Arms: Continuous catheter drainage
Drug: Conservative treatment — Including antibiotics,somatostatin, proton pump inhibitors and sufficient fluid resuscitation
  Arms: Conservative treatment

SUMMARY:
Acute fluid collections is common in patients with severe acute pancreatitis (SAP). But the treatment for this is controversial. In this study, the investigators aim to evaluate the different effects of three different treatment protocols which is repeated aspiration, continuous catheter drainage and conservative treatment. The investigators suppose repeated aspiration could not only solve acute fluid collections, but also lower the rate of pancreatic infection.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms and signs of acute pancreatitis according to Atlanta criteria and if pancreatic or/and peripancreatic fluid collections were confirmed by ultrasound and computed tomography examination
* CT density < 30Hu
* Within 7 days from the onset of the disease
* Available approach for percutaneous penetrate

Exclusion Criteria:

* Pregnant pancreatitis
* Receiving surgery or aspiration before;need of early surgery
* Infected fluid collection

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Estimated)
Dates: Start 2011-01; Primary Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
pancreatic infection | 28 days
mortality | 28 days

SECONDARY OUTCOMES:
inflammation parameters | 28 days
intra abdominal pressure | 28 days
complications | 28 days
  intestinal fistula , major bleeding, etc.
ICU duration | day one until discharge
hospital duration | day one until discharge
SIRS | 28 days
MODS | 28 days

CONTACTS AND LOCATIONS:
Locations (1):
- Department of SICU, Research Institute of General Surgery Jinling Hospital,, Nanjing, Jiangsu, China